CLINICAL TRIAL: NCT03795896
Title: Ocular Ultrasonography in Assessing Severity and Management of Increased Intracranial Pressure in Traumatic Brain Injury
Brief Title: Ocular Ultrasonography as a Tool for Monitoring the Management of Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Abdelraouf Elsharkawy, Lecturer of anesthesia and surgical intensive care, Mansoura University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ms/15.05.88
Record Dates: First submitted 2019-01-01; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: prospective observational study
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optic nerve sheath diameter (Experimental): The intracranial pressure will be measured by optic nerve sheath diameter while the patient in supine position with 30 -degree bed position .The linear probe in the two -dimensional mode will be placed gently on the upper eyelid without pressure .In linear horizontal orientation for both right and left optic nerve sheath will be measured
  Interventions: Diagnostic Test: Optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter — The intracranial pressure will be measured by the optic nerve sheath diameter and after giving the mannitol osmotherapy the intracranial pressure will be monitored by the optic nerve sheath diameter
  Other Names: ONSD

SUMMARY:
Raised intracranial pressure (ICP) is a common and life threatening condition especially in patients with traumatic brain injury.There are many methods for monitoring the increased (ICP) either invasive or non- invasive ,but the gold standard is invasive method. Optic nerve sheath ultrasonography provides a very promising bedside tool for detection of increased ICP. This study will monitor the dynamic changes of intracranial pressure by optic nerve sheath diameter (ONSD) in response to mannitol osmotherapy

DETAILED DESCRIPTION:
Traumatic brain injury is the main cause of increased intracranial pressure (ICP) in the intensive care .

There are multiple methods for monitoring the raised ICP either invasive or non-invasive.The gold standard is the invasive devices because it is more accurate and reliable .However ,it requires a surgical intervention which has many hazards such as (infection ,hemorrhage,malfunction ).

Optic nerve sheath ultrasonography is a promising bedside tool for detection of increased ICP. The optic nerve is surrounded by cerebro-spinal fluid ,thus if the circulation of cerebro-spinal fluid not blocked ,an increase in ICP will be transmitted through the subarachnoid space around the optic nerve within the nerve sheath especially the retro-bulbar segment.

The study will be conducted to monitor the dynamic changes of intracranial pressure by optic nerve sheath diameter (ONSD) in response to mannitol osmotherapy as a primary outcome and secondary to evaluate the efficacy of ONSD in assessing the severity of the disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic brain injury

Exclusion Criteria:

* Patients with history of optic neuritis
* past history of eye trauma
* patient with optic nerve trauma
* patient with history of arachnoid cyst of the optic nerve
* high myopic patients
* patients with cavernous sius mass

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the changes in the intracranial pressure | from 20 minutes before mannitol therapy (basal reading) till 48 hours after the end of mannitol infusion
  It will be monitored and recorded the changes in intracranial pressure to the mannitol therapy .Basal (before mannitol therapy).20 minutes after the end of mannitol infusion ,2 hours ,6 hours,12 hours ,24 hours and 48 hours after the end of mannitol infusion

SECONDARY OUTCOMES:
Assessing the changes in the heart rate | from 20 minutes before mannitol therapy (basal reading ) till 48 hours after the end of mannitol infusion
  It will be recorded basal (before mannitol therapy).20 minutes after the end of mannitol infusion ,2 hours ,6 hours,12 hours ,24 hours and 48 hours after the end of mannitol infusion
Assessing the changes in the mean arterial pressure | from 20 minutes before mannitol therapy(basal reading) till 48 hours after the end of mannitol infusion
  It will be calculated according to the formula systolic blood pressure+2(diastolic blood pressure)recorded basal (before mannitol therapy).20 minutes after the end of mannitol infusion ,2 hours ,6 hours,12 hours ,24 hours and 48 hours after the end of mannitol infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Reem Abdelraouf Elsharkawy, Al Mansurah, Dakahlia Governorate, Egypt